CLINICAL TRIAL: NCT00681616
Title: Randomized Clinical Trial of Tissue Ultrafiltration and Pressure Monitoring for the Diagnosis and Prevention of Compartment Syndrome
Brief Title: Study of New Catheter & Pressure Monitor System to Help Prevent Compartment Syndrome From Developing in the Injured Leg
Acronym: TS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Twin Star Medical, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Janelle Antil, Director, Clinical Affairs, Twin Star Medical, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GE-4073; DoD Proposal:06275001; Award #:W81XWH-07-1-0243
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-02

CONDITIONS: Compartment Syndrome
Keywords: Anterior compartment syndrome; Tibia; Trauma; Blood circulation; Nerve compression syndromes
MeSH Terms: conditions — Compartment Syndromes; Anterior Compartment Syndrome; Wounds and Injuries; Nerve Compression Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Compartment Monitoring System with Active Fluid Removal
  Interventions: Device: Compartment Monitoring System (CMS); Device: Compartment Monitoring System with Active Fluid Removal
- 2 (Active Comparator): Compartment Monitoring System (CMS) without fluid removal
  Interventions: Device: Compartment Monitoring System (CMS); Device: Compartment Monitoring System without fluid removal

INTERVENTIONS:
Device: Compartment Monitoring System (CMS) — The CMS consists of an Introducer, Pressure Measurement & Fluid Collection (PMFC) catheter, a Fluid Collection (FC) catheter and Compartment Pressure Monitor. The PMFC catheter removes fluid and monitors pressure via a solid-state fiber optic transducer at the tip of the catheter. The FC catheter only removes fluid and does not have a pressure transducer at the tip. The CMS Monitor senses, displays and records compartment pressure as measured by up to two PMFC catheters. In addition, the CMS Monitor measures subject blood pressure using a provided cuff for calculating the perfusion pressure of the muscle compartment.
  Other Names: Twin Star Monitor; Twin Star Catheters
Device: Compartment Monitoring System with Active Fluid Removal — Compartment Monitoring System with Active Fluid Removal
  Other Names: Twin Star Monitor; Twin Star Catheters
  Arms: 1
Device: Compartment Monitoring System without fluid removal — Compartment Monitoring System without fluid removal
  Other Names: Twin Star Monitor; Twin Star Catheters
  Arms: 2

SUMMARY:
An investigation of a new catheter and pressure monitor system that may help to prevent a complication called compartment syndrome from developing in an injured leg. Compartment syndrome occurs when too much fluid builds up in the muscles of the injured leg. This causes a lot of swelling and increases pressures within the leg that can cause permanent damage muscles and nerves in the leg.

DETAILED DESCRIPTION:
Compartment Syndrome (CS) may occur in patients with a fracture or crushing injury to an extremity. The current standard-of-care for patients at risk of developing CS is clinical by watching for signs and symptoms of CS, and if needed, measuring the pressure within the muscle compartment (intramuscular pressure, IMP). Currently, IMP measurements are made by placing a percutaneous pressure sensor into the targeted muscle compartment, which is then attached to a pressure monitor. Whenever the clinical exam and/or pressure measurements suggest that CS is developing, fasciotomy is generally performed immediately.

Twin Star Medical has developed a novel Compartment Monitoring System (CMS) that consists of a pressure monitoring module and two types of catheters. Both Twin Star Catheters remove interstitial tissue fluid, which may contribute to a reduction in compartment pressure, and which may be used for clinical analysis to determine if certain analyte indicators of muscle injury (biomarkers) can be predictive of CS development. One type of catheter Pressure Measurement/Fluid Collection, (PMFC), removes fluid and monitors pressure via a solid-state fiber optic transducer at the tip of the catheter. The other type of catheter, Fluid Collection (FC), only removes fluid and does not have a pressure transducer at the tip. The monitoring module senses, displays and records pressure as measured by the PMFC catheter as well as provides a vacuum source, which is required for the operation of the fluid removal catheter. The Twin Star CMS Monitoring Module has been successfully tested to (1) ensure the delivery of the specified functional performance requirements needed to reliably operate the Twin Star Catheter, and (2) meet current electrical safety standards established for clinical use. The first model of the Twin Star catheter and monitor was reviewed and approved by the Food and Drug Administration (FDA) for the indications of pressure measurement and the withdrawal of interstitial fluid. The devices being used for this clinical study represent the newly designed catheter and monitor and are not FDA approved and are therefore considered investigational. It is anticipated that the second-generation model of the catheter and monitor will be submitted to the FDA for approval while this study is being conducted.

The purpose of this Study is to determine if the removal of interstitial fluid by the Twin Star Catheter can lower muscle compartment pressure and impact other measures of subject clinical status, including possible reduction of the need for fasciotomy. The Study population will be Subjects who have suffered an isolated tibial fracture (open or closed) requiring surgical stabilization within 72 hours of injury. This Study will use an Adaptive study design in which a total of up to 90 subjects will be enrolled. All Subjects will receive the Twin Star catheters, which will be inserted at the end of the surgical procedure to stabilize the tibia fracture and will be connected to the pressure monitor before leaving the surgical room. The catheters will be used for the first 24-hours after surgical fixation of the affected lower leg in order to (1) measure and record muscle compartment pressure, and (2) remove accumulated interstitial fluid in the subset of subjects that are randomized to the Treatment Group. The first 20 Subjects (Phase 1) will not be randomized; all will be actively treated but with different combinations of catheters and vacuum levels. The purpose of Phase I of the study is to optimize treatment parameters that will be used in the remaining 70 subjects, which will constitute Phase II. All subjects will receive a total of 3 catheters placed in the anterior compartment. Subjects in Phase 1 will be enrolled into two groups: 1) receiving constant vacuum (-150 mmHg) and fluid removal or, 2) receiving intermittent vacuum (-50 mmHg) and fluid removal. Within the anterior compartment, there will be one PMFC and 2 FC catheters inserted.

The first 10 subjects in Phase 1 will all be treated with single-fiber catheters, but with one of two different vacuum levels (intermittent at -50 mmHg or constant at -150 mmHg). After the first 10 subjects have completed the study, fluid removal results will be analyzed. If results demonstrate that fluid in the anterior compartment is being withdrawn at a rate of ≥ 0.5 mls/24 hours, the second group of 10 subjects will continue using the same single fiber catheters. If the results of the first 10 subjects demonstrate fluid is being withdrawn in the anterior compartment at < 0.5 mls/24 hours, the next 10 subjects will instead receive treatment with two multi-fiber FC catheters plus the same PMFC catheter.

After the first 20 subjects have been enrolled in the study, the remaining subjects to be enrolled in Phase 2 will be randomized to either a Treatment or Control group. Both groups will receive treatment with whichever combination of catheter type (single or multi-fiber) and vacuum (constant or intermittent) was most efficacious in terms of fluid removal in Phase 1. The randomization will determine whether subjects will receive no vacuum at all (Control Group: Monitoring alone) or the fluid removal mode that was shown to be best in the first phase of the study (Treatment Group: Monitoring plus Fluid Removal).

The rationale for the adaptive study design is that we have developed second-generation catheters whose fluid removal function has not been optimized in vivo in humans. Although our first generation catheter used multi-fibers, animal study results have demonstrated that single-fiber catheters remove the same amount of fluid in vivo as multi-fiber catheters, but can be made much smaller than multi-fiber catheters.

The Subject's length of initial hospital stay will be determined by the attending physician based on the subject's medical condition(s). The standard-of-care for routine clinical compartment pressure monitoring will apply to both the vacuum and non-vacuum groups in this Study with the catheters being left in place for 24 hours. Compartment syndrome is a dignosis that depends on clinical assessment supplemented by pressure measurement. Throughout the study, the treating physicians will monitor the subjects according to standard clinical practice and will apply standard clinical judgment regarding the diagnosis of compartment syndrome. Treating physicians may end the study and perform fasciotomy if they feel it is necessary because of clinical suspicion that compartment syndrome is developing. A two-week and a 3-month follow-up visit will be required post discharge, coinciding with typical clinical follow-up visits. The purpose of the two-week visit will be primarily to assess whether there have been any adverse consequences related to the catheter. The purpose of the three-month assessment will be primarily to look for any evidence of the sequelae of missed or untreated compartment syndrome, such as clawing of the toes or persistent neurologic dysfunction. Functional outcomes will be measured during these follow-up visits as well as the occurrence of any adverse events since discharge. Functional outcomes will include an assessment of whether any loss of motor function resulted as part of the primary injury.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a tibial shaft fracture requiring intramedullary nailing or bicondylar tibial plateau fracture requiring application of a knee-spanning external fixator.
* Operative procedure (nailing or external fixation) performed within 72 hours of injury.
* The Subject is between 18 and 60 years of age.
* Able to understand what he/she is being asked to do, willing/able to understand and sign the Informed Consent to return for follow-up visits at 2 weeks and 3 months post surgery.

Exclusion Criteria:

* Current evidence of CS prior to Study.
* Surgical stabilization will result in the presence of a bead pouch or wound vac or other dressing that would interfere with placement of any of the three Catheters in the anterior compartment.
* The Subject has a medical condition(s) that precludes use of Catheters, such as dermatologic conditions, immunological deficits or traumatic skin lesions that interfere with Catheter placement.
* The Subject has co-morbidities that may place the Subject at risk of hypotension (e.g., significant blood loss, heart failure, significant chest or abdominal trauma, septicemia, pelvic fractures, femur fractures or massive soft tissue trauma.)
* Likely problems, in the investigator's judgment, with maintaining follow-up (including developmental delay, address greater than 2 hours drive from the treating institution, substance abuse problems, intoxication, current or pending incarceration, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To determine if use of Twin Star catheter with active fluid removal reduces muscle compartment pressure vs Twin Star catheter without fluid removal by comparing the randomized groups. Success will be defined by a p-value less than 0.05 (two-sided). | fluid removal will be collected & recorded at 2, 4, 8, 16, & 24 hrs after catether insertion.

SECONDARY OUTCOMES:
Compares the treatment and control groups on change in perfusion pressure (defined as diastolic blood pressure minus IMP) over time. The randomized groups will be compared with a two-sided p-value less than 0.05 defining success. | Perfusion pressure will be collected and recorded at 2, 4, 8, 16 & 24 hrs post-catheter insertion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schmidt, MD, Principal Investigator — Hennepin County Medical Center (HCMC); Janelle M Antil, Study Director — Twin Star Medical, Inc.
Locations (13):
- United States (13):
  - University of California, Irvine Medical Center, Orange, California
  - University of California - San Francisco / San Franciso General Hospital, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - Loyola University Medical Center, Maywood, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Washington University Orthopedics, St Louis, Missouri
  - ECMC - SUNY Buffalo, Buffalo, New York
  - Ohio State University, Columbus, Ohio
  - University of Tennessee/Campbell Clinic-InMotion Musculoskeletal Institute, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Background] Blick SS, Brumback RJ, Poka A, Burgess AR, Ebraheim NA. Compartment syndrome in open tibial fractures. J Bone Joint Surg Am. 1986 Dec;68(9):1348-53. PMID 3782206
- [Background] Hargens AR, Akeson WH, Mubarak SJ, Owen CA, Evans KL, Garetto LP, Gonsalves MR, Schmidt DA. Fluid balance within the canine anterolateral compartment and its relationship to compartment syndromes. J Bone Joint Surg Am. 1978 Jun;60(4):499-505. PMID 670272
- [Background] Hargens AR, Schmidt DA, Evans KL, Gonsalves MR, Cologne JB, Garfin SR, Mubarak SJ, Hagan PL, Akeson WH. Quantitation of skeletal-muscle necrosis in a model compartment syndrome. J Bone Joint Surg Am. 1981 Apr;63(4):631-6. PMID 7217130
- [Background] Heppenstall RB, Scott R, Sapega A, Park YS, Chance B. A comparative study of the tolerance of skeletal muscle to ischemia. Tourniquet application compared with acute compartment syndrome. J Bone Joint Surg Am. 1986 Jul;68(6):820-8. PMID 3733772
- [Background] Janzing HM, Broos PL. Routine monitoring of compartment pressure in patients with tibial fractures: Beware of overtreatment! Injury. 2001 Jun;32(5):415-21. doi: 10.1016/s0020-1383(01)00005-5. PMID 11382429
- [Background] Schmidt AH, Tvedte E. The Financial Implications of Compartment Syndrome. Poster, American Academy of Orthopaedic Surgeons Annual Meeting, San Diego, CA, Feb 13-18, 2007.
- [Background] Tornetta P 3rd, Templeman D. Compartment syndrome associated with tibial fracture. Instr Course Lect. 1997;46:303-8. No abstract available. PMID 9143975
- [Background] Woll TS, Duwelius PJ. The segmental tibial fracture. Clin Orthop Relat Res. 1992 Aug;(281):204-7. PMID 1499212